CLINICAL TRIAL: NCT05077696
Title: Contribution of the Neurofilament Assay for the Diagnosis of ALS (Amyotrophic Lateral Sclerosis) in Situations of Diagnostic Standoff After Evaluation in an Expert ALS Center
Brief Title: Neurofilament Assay for the Diagnosis of ALS
Acronym: FILSLAN-NF
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP210917; 2021-A02460-41 (Other: IDRCB)
Record Dates: First submitted 2021-10-01; First posted 2021-10-14 (Actual); Last update posted 2021-10-14 (Actual); Status verified 2021-09

CONDITIONS: Progressive Motor Neuron Disease Without Definite Diagnosis
Keywords: ALS; Neurofilaments; NFL; pNFH; Amyotrophic Lateral Sclerosis; progressive motor neuron disease
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with progressive motor neuron disease without definite diagnosis: Patients with progressive motor neuron disease without definite diagnosis
  Interventions: Other: Drawing a tube of blood (serum)

INTERVENTIONS:
Other: Drawing a tube of blood (serum) — dosage of neurofilaments and comparison with a final diagnosis one year after sampling.

SUMMARY:
The aim of the study is to evaluate the interest of the determination of pNFH and NFL neurofilaments in serum for the diagnosis of ALS in patients with a diagnostic standoff after evaluation in an expert ALS center. The hypothesis is that one of these biomarkers, or their combined analysis, will make it possible to confirm or invalidate the diagnosis of ALS.

DETAILED DESCRIPTION:
For this study, which aims to evaluate a test to help in the diagnosis of ALS that could be integrated into routine practice, it was preferred to use blood tests. Blood sampling is significantly less invasive than CSF sampling, and more easily generalized, including in ambulatory conditions.

ELIGIBILITY:
Inclusion criteria :

Subjects with first and/or second motor neuron disease, evolving clinically and/or electrically over at least 12 months, not meeting the diagnostic criteria for ALS (revised El Escorial criteria):

* Isolated peripheral motor neuron disease (at least one region of the PNM) OR
* Isolated central motor neuron involvement (at least two areas of the MNC) OR
* associated involvement of the MNP and MNC but in the presence of an associated pathology responsible for a persistent diagnostic doubt (double narrow cervical and lumbar canal, associated evolving cancer evoking a paraneoplastic syndrome without specific antibody found) Age superior to 18 years Management and follow-up in one of the French ALS centers Patient able to express his non-opposition Affiliation with social security or beneficiary of such a plan

Non-inclusion criteria:

Refusal of the patient Person under a legal protection measure (guardianship, curatorship or safeguard of justice).

Person deprived of liberty by judicial or administrative decision.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with progressive motor neuron disease without a definite diagnosis.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-11-01 (Estimated); Primary Completion 2023-11-01 (Estimated); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
contribution of pNFH and NFL neurofilaments assays | 1 year
  contribution of pNFH and NFL neurofilaments assays in serum for the positive diagnosis of ALS in a selected population of patients with progressive motor neuron disease without definite diagnosis

SECONDARY OUTCOMES:
Value of the combined pNFH and NFL neurofilament assay in serum versus the pNFH and NFL assay alone | 1 year
  To evaluate the value of the combined pNFH and NFL neurofilament assay in serum versus the pNFH and NFL assay alone for the positive diagnosis of ALS in a selected population of patients with progressive motor neuron disease without a definite diagnosis.